CLINICAL TRIAL: NCT05706259
Title: A Comparative Vitamin D Bioavailability Study Following Supplementation of an Orodispersible, Chewable Tablet and Soft Gelatin Capsule Vitamin D3 Supplementation in Vitamin D Deficient Healthy Adults
Brief Title: A Comparative Dissolution and Absorption Study of an Orodispersible Powder, Chewable Tablet and Soft Gel Capsule Vitamin D3 Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No. LUMHS/REC/-152
Record Dates: First submitted 2023-01-11; First posted 2023-01-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soft gelatin vit D supplement (Active Comparator): In this arm subjects will receive a weekly single dose 200000 IU soft gelatin capsule of vitamin D3 for 3-weeks
  Interventions: Dietary Supplement: Soft gelatin 200000 IU vitamin D3 capsule
- Orodispersible vit D supplement (Experimental): In this arm subjects will receive a weekly single dose 200000 IU orodispersible (sachet) vitamin D3 for 3-weeks
  Interventions: Dietary Supplement: Orodispersible (sachet) 200000 IU vitamin D3

INTERVENTIONS:
Dietary Supplement: Soft gelatin 200000 IU vitamin D3 capsule — Weekly single dose for 3-weeks
  Arms: Soft gelatin vit D supplement
Dietary Supplement: Orodispersible (sachet) 200000 IU vitamin D3 — Weekly single dose for 3-weeks
  Arms: Orodispersible vit D supplement

SUMMARY:
This is an open-labelled, randomized controlled clinical trial aimed to compare the pharmacokinetics of an orodispersible vs a soft gelatin vitamin supplementation in vitamin D deficient healthy adults.

DETAILED DESCRIPTION:
Vitamin D is a fat-soluble vitamin used by the body for normal bone development and maintenance by increasing the absorption of calcium, magnesium, and phosphate. Vitamin D also plays a role in the nervous system, musculoskeletal system and immune system. Vitamin D deficiency has been linked with diverse health conditions including diabetes, cardiovascular diseases, breast, colorectal and prostate cancer, dementia, depression, erectile dysfunction, osteoporosis, and bone disorders. Vitamin D deficiency is a global healthcare challenge. To overcome vitamin D deficiency, a daily vitamin D supplementation of 200-1000 IU or a high dosage from 25000 to 200000 IU for 4-6 weeks, is normally recommended.

Vitamin D supplements are available over the counter in different delivery vehicles (formulations) to reach the circulatory system. In the present study the investigators aim to evaluate the pharmacokinetics of an orodispersible vitamin D supplement vs a conventional oral soft gelatin capsule, in vitamin D deficient healthy adults to assess how different vitamin D supplement formulations can efficiently overcome the vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults aged 18 - 60 years
* Vitamin D deficiency as shown by serum levels of 25 (OH) D3 levels of < 20 ng/mL
* Able to provide informed written consent

Exclusion Criteria:

* Clinically significant abnormal laboratory parameters (such as complete blood count, CRP, d-dimer, liver enzymes, creatinine) indicative of physical illness, especially hypercalcemia and hypercalciuria
* History of hypersensitivity to vitamin D3 supplements
* History of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine, or neurological diseases
* Prior use of medications in general containing calcium, magnesium, or vitamin D3, four weeks before the start of the study
* Participation in the evaluation of any investigational product or blood donations in the last three months before this study
* Any other significant disease or disorder that, in the opinion of the Physician, may either put the participant at risk because of participation in the study, or may influence the results of the study, or the participant's ability to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in serum level of 25 (OH) D | 6 weeks
  Effect on the vitamin D deficiency level

SECONDARY OUTCOMES:
Effect on liver enzymes profile | 6 weeks
  Change in serum Alanine transaminase (ALT) level
Effect on liver enzymes profile | 6 weeks
  Change in serum Aspartate transaminase (AST) level
Effect on liver enzymes profile | 12 weeks
  Change in serum Aspartate transaminase (AST) level
Effect on liver enzymes profile | 6 weeks
  Change in serum Albumin level
Effect on liver enzymes profile | 6 weeks
  Change in serum Billirubin level
Effect on liver enzymes profile | 6 weeks
  Change in serum Gamma-glutamyltransferase (GGT) level
Effect on kidney function | 6 weeks
  Change in serum creatinine level

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat Medical University Hospital, Jamshoro, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bano A, Abrar S, Brilli E, Tarantino G, Bugti AA, Fabbrini M, Conti G, Turroni S, Bugti M, Afridi F, Mureed S, Zada H, Din Ujjan I, Ashraf S, Ghafoor A, Khan S, Khan A. A comparative absorption study of sucrosomial(R) orodispersible vitamin D3 supplementation vs. a reference chewable tablet and soft gel capsule vitamin D3 in improving circulatory 25(OH)D levels in healthy adults with vitamin D deficiency-Results from a prospective randomized clinical trial. Front Nutr. 2023 Aug 17;10:1221685. doi: 10.3389/fnut.2023.1221685. eCollection 2023. PMID 37662595